CLINICAL TRIAL: NCT03998345
Title: A First-in-Human, Open-label, Phase 1 Dose-Escalation Study of 609A in Subjects With Locally Advanced/Metastatic Solid Tumors in China
Brief Title: Phase 1, First in Human, Open-Label, Dose-Escalation Study of 609A in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-609-UND-I-01
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 609A group (Experimental): Dose escalation will be conducted using a traditional 3+3 design. Dose Escalation Level cohort 1. Dose 1 mg/kg, Q3W, IV. Subjects 3-6； Dose Escalation Level cohort 2. Dose 3 mg/kg, Q3W, IV. Subjects 3-6； Dose Escalation Level cohort 3. Dose 200mg, Q3W, IV. Subjects 3-6； Dose Escalation Level cohort 4. Dose 10 mg/kg, Q3W, IV. Subjects 3-6. If 10mg/kg cannot be tolerated, add a dose level of 400mg to assess the tolerance
  Interventions: Drug: 609A

INTERVENTIONS:
Drug: 609A — 609A is a recombinant anti-PD-1 humanized IgG4 kappa antibody that targets the human PD-1

SUMMARY:
Phase 1, First in Human, Open-Label, Dose-Escalation Study of 609A in the Patients with Locally advanced/Metastatic Solid Tumors in China.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), open-label, phase 1 dose-escalation study of 609A in China, a recombinant monoclonal anti-PD-1 antibody product, in subjects with Locally advanced/Metastatic Solid Tumors, who must have failed standard treatment (disease progression or intolerance) or lack of standard treatment. If there is a driver gene variant, the subjects must have failed the standard treatment for the driver gene, and there is no other standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible for participation in this study:

* Able to understand and willing to sign the Informed Consent Form(ICF).
* No limit gender .
* Age range: from 18 years to 70 years.
* Subjects with histologically or cytologically confirmed locally advanced-stage or metastatic tumor must have failed standard treatment (disease progression or intolerance) or lack of standard treatment. If there is a driver gene variant, the subjects must have failed the standard treatment for the driver gene, and there is no other standard treatment.
* Patients who had been previously treated for brain metastases, must have asymptomatic or radiographic/clinical stability and no need for steroid therapy of brain metastases to be enrolled in this study within 4 weeks prior to enrollment .
* According to RECIST1.1, Patients must have at least one measurable lesion (target or non-target).
* ECOG scores 0,1 or 2.
* Life expectancy ≥3 months
* Must have adequate organ function, prior to start of 609A, including the following:

  1. Bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.0 ×109/L; platelet count≥ 100 × 109/L; hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L;
  2. Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 3 × ULN (≤5 × ULN if with liverinvolvement)
  3. Renal: serum creatinine ≤1.5 times the ULN or estimated creatinineclearance ≥50mL/min (Cockroft and Gault formula).
  4. Coagulation tests INR≤ 2 (Exception: INR 2 to ≤ 3 is acceptable for subjects on Warfarin anticoagulation), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Female patient with fertility or male patient whose partner has fertility should use one or more contraceptive methods for contraception from the screening period to five half-lives after the last treatment. These measures include, but are not limited to, oral or implantable injections of hormonal contraceptives; intrauterine birth control ring or placement of intrauterine system (IUS) hormone-releasing intrauterine device; or use of barrier methods such as condoms or septum and spermicide products. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to the first dose of study drug. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled:

* History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or excipients in 609A drug formulation.
* Subjects who had experienced severe allergic reactions after administration of other monoclonal antibodies
* Pregnant or nursing females
* Regarding previous anti-tumor therapy:

  1. Subjects who have received any anticancer drugs approved or investigational, including chemotherapy,hormonal therapy (Exceptions: hormone-replacement therapy, testosterone or oral contraceptives), biologic therapy, have stopped treatment for less than 3 weeks or 5 half-lives, whichever is longer, before first dose of 609A.
  2. Subjects who have stopped systemic radiation therapy less than 3 weeks before first dose of 609A, or local radiotherapy or radiation therapy for bone metastases less than 2 weeks before first dose of 609A. Therapeutic radiopharmaceuticals were taken within 8 weeks before first dose of 609A.
  3. Subjects who have received prior immunotherapies targeting T cell stimulation such as (e.g. anti-PD-1, anti- PD-L1 or anti-CTLA-4) ,have stopped treatment less than 3 months before first dose of 609A.
  4. The ADA antibody of anti-PD-1 drug in plasma was positive during screening.
  5. Subjects who have received immunogonists (such as interleukin-2 gamma interferon, oncolytic virus, mistletoe extract, etc.) or drugs known to interfere with major organ function (e.g., hypericin) , have stopped treatment less than 4 weeks or 5 half-lives, whichever is longer, before first dose of 609A.
* Subjects with severe chronic or active infections requiring systemic antimicrobial, antifungal, or antiviral treatment, including tuberculosis.
* HIV infection
* Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer< 1000 cps/mL or 200 IU/mL) or cured Hepatitis C (negative HCV RNA test) may been rolled
* Subjects with history of interstitial lung disease or noncommunicable pneumonia, or uncontrolled pulmonary fibrosis or acute pulmonary disease . Local interstitial pneumonia due to radiotherapy was excluded.
* Acute or chronic uncontrolled renal disease( Exception: Renal carcinoma, metastatic renal cancer), pancreatitis or liver disease (per investigator assessment).
* Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5. 0, with exception of the residual hair loss.
* Any SAE occurred during previous pd-1 / pd-l1 treatment, including but not limited to interstitial pneumonia and myocarditis.
* Subjects who experienced immunotherapy-related adverse events (irAE) grade ≥ 3, or who had to discontinue prior anti-PD-1, anti-PD-L1, or CTL4 treatment due to irAEs of any grade
* Subjects with acute myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack occurred within 6 months prior to admission. Subjects with congestive heart failure rated as grade 2 or above (including grade 2) by the New York college of cardiology (NYHA) ,LVEF<50%.And subjects with the following heart diseases:

  1. ECG QTcF> 480 msec during screening.
  2. Right bundle branch block and left anterior half branch block or complete left bundle branch block.
  3. Subjects with congenital long QT syndrome or a family history of unexpected sudden cardiac death.
  4. Subjects with ventricular tachyarrhythmia or history of tachyarrhythmia.
  5. Bradycardia with obvious clinical significance (< 50 times/min).
  6. Subjects using pacemakers.
  7. Subjects with other heart disease with significant clinical significance.
* Sustained systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg after antihypertensive medication.
* Fever and neutropenia occurred within 1 week before the first dose of 609A.
* Subjects who have had major surgery within 21 days before the first dose of 609A ((excluding diagnostic biopsies).
* Live attenuated vaccines were administered within 28 days before the first dose of 609A.
* Patients who had received treatment with any herbal or alternative therapies or Chinese prepared medicine within 7 days before the first dose of 609A.
* History of primary immunodeficiency, stem cell or organ transplant, or previous clinical diagnosis of tuberculosis disease.
* Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded; these include but are not limited to subjects with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain- Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, hepatitis, toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or antiphospholipid syndrome.
* Subjects with condition requiring systemic treatment with either corticosteroids (>15 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the planned first dose of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Ophthalmologic, nasal and intra-articular injections of steroids are acceptable.
* Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of clotting disorders), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications.
* Any other conditions not suitable for subjects to be enrolled in this study, as determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-12-24 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | for 90 days
  To access adverse events (AEs) per the NCI CTCAE 5.0.
The MTD | for 90 days
  Maximum Tolerated Dose， if any, and RP2D (s) for 609A will be determined.

SECONDARY OUTCOMES:
AUC | for 90 days
  Area Under the Curve of 609A
Cmax | for 90 days
  Maximum Plasma Concentration of 609A
t1/2 | for 90 days
  Half life of 609A in blood
CL | for 90 days
  Plasma clearance of 609A
ORR | for 1 year
  the rate of completely response [CR] and partial response [PR] patients
DCR | for 1 year
  disease control rates of the patients with 609A
DOR | for 1 year
  Duration of response of the patients with 609A
PFS | for 1 year
  Progression-free survival of the patients with 609A
OS | for 1 year
  overall survival of the patients with 609A
ADA | for 1 year
  to detect the presence of anti-609A antibody
PD-L1 | for 1 year
  to evaluate the expression of pd-l1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Chinese academy of medical sceience, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided